CLINICAL TRIAL: NCT03172494
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide, Insulin Degludec, and Liraglutide in Chinese Subjects With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetic Drugs (OADs)
Brief Title: A Trial Comparing Insulin Degludec/Liraglutide, Insulin Degludec, and Liraglutide in Chinese Subjects With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetic Drugs (OADs)
Acronym: DUAL™ I China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4148; U1111-1154-6671 (Other: World Health Organization (WHO)); CTR20170004 (Registry Identifier: China Drug Trials (China))
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Insulin degludec/liraglutide (Experimental)
  Interventions: Drug: Insulin degludec/liraglutide
- Insulin degludec (Active Comparator)
  Interventions: Drug: Insulin degludec
- Liraglutide (Active Comparator)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Insulin degludec/liraglutide — Subcutaneously (s.c., under the skin)administration once daily in combination with metformin.
  For 26 weeks.
  Arms: Insulin degludec/liraglutide
Drug: Insulin degludec — Subcutaneously (s.c., under the skin)administration once daily in combination with metformin.
  For 26 weeks.
  Arms: Insulin degludec
Drug: Liraglutide — Subcutaneously (s.c., under the skin)administration once daily in combination with metformin.
  For 26 weeks.
  Arms: Liraglutide

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to confirm the efficacy of insulin degludec/liraglutide in controlling glycaemia in Chinese subjects with type 2 diabetes mellitus inadequately controlled on oral antidiabetic agents

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Type 2 diabetes mellitus (clinically diagnosed)
* Male or female, age at least 18 years at the time of signing informed consent
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis, with the aim of a median of8.3%. When approximately 50% of the randomised subjects have an HbA1c above 8.3%, the remaining subjects randomised must have an HbA1c below or equal to 8.3%; or when approximately 50% of the randomised subjects have an HbA1c below or equal to 8.3%, the remaining subjects randomised must have an HbA1c above 8.3%
* Current treatment for at least 90 calendar days prior to screening with metformin plus/minus one other OAD: α-glucosidase inhibitors, sulphonylureas, glinides or thiazolidinediones. For above or equal to 60 calendar days prior to screening subjects should be on a stable dose of:
* Metformin (above or equal to 1500 mg or max tolerated dose) or
* Metformin (above or equal to 1500 mg or max tolerated dose) and sulphonylureas (above or equal to half of the max approved dose according to local label) or
* Metformin (above or equal to 1500 mg or max tolerated dose) and glinides (above or equal to half of the max approved dose according to local label) or
* Metformin (above or equal to 1500 mg or max tolerated dose) and α-glucosidase inhibitors (above or equal to half of the max approved dose according to local label) or
* Metformin (above or equal to 1500 mg or max tolerated dose) and thiazolidinediones (above or equal to half of the max approved dose according to local label)

Exclusion Criteria:

* Treatment with insulin (except for short-term treatment at the discretion of the investigator)
* Treatment with glucagon-like-peptide-1 receptor agonists or dipeptidyl-peptidase-4 inhibitors within 90 days prior to screening
* Impaired liver function, defined as alanine aminotransferase above or equal to 2.5 times upper normal range
* Impaired renal function defined as serum-creatinine above or equal to 133 μmol/L for males and above or equal to 125 μmol/L for females, or as defined according to local contraindications for metformin
* Screening calcitonin above or equal to 50 ng/L
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
* Cardiac disorder defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the last 12 months prior to screening and/or planned coronary, carotid or peripheral artery revascularisation procedures
* Severe uncontrolled treated or untreated hypertension (systolic blood pressure above or equal to 180 mmHg or diastolic blood pressure above or equal to 100 mmHg
* Proliferative retinopathy or maculopathy (macular oedema), requiring acute treatment
* History of pancreatitis (acute or chronic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (22):
- China (22):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Cangzhou, Hebei
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Changzhou, Jiangsu
  - Novo Nordisk Investigational Site, Huai'an, Jiangsu
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Yinchuan, Ningxia
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Jinan, Shandong
  - Novo Nordisk Investigational Site, Pudong New District, Shanghai Municipality
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
  - Novo Nordisk Investigational Site, Fuzhou

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wang W, Agner BFR, Luo B, Liu L, Liu M, Peng Y, Qu S, Stachlewska KA, Wang G, Yuan G, Zhang Q, Ning G. DUAL I China: Improved glycemic control with IDegLira versus its individual components in a randomized trial with Chinese participants with type 2 diabetes uncontrolled on oral antidiabetic drugs. J Diabetes. 2022 Jun;14(6):401-413. doi: 10.1111/1753-0407.13286. PMID 35762390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 38 sites in China mainland.
Pre-assignment Details: Participants were randomised in a 2:1:1 manner to receive insulin degludec/liraglutide, insulin degludec or liraglutide in combination with metformin.
Groups:
- Insulin Degludec/Liraglutide: Participants were to receive Insulin degludec/liraglutide subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 10 dose steps (10 units insulin degludec and 0.36 milligrams (mg) liraglutide) initially. The dose was then adjusted twice weekly based on pre-breakfast self-measured plasma glucose (SMPG) target of 4.0-5.0 millimoles/litre (mmol/L). The maximum dose was 50 dose steps (50 units insulin degludec and 1.8 mg liraglutide). One dose step corresponded to 1 unit insulin degludec per 0.036 mg liraglutide.
- Insulin Degludec: Participants were to receive Insulin degludec subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 10 units insulin degludec initially. The dose was then adjusted twice weekly based on pre-breakfast SMPG target of 4.0-5.0 mmol/L. There was no maximum dose for Insulin degludec.
- Liraglutide: Participants were to receive liraglutide subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 0.6 mg initially. The dose was then escalated in weekly increments of 0.6 mg to reach a target dose of 1.8 mg. Liraglutide dose of 1.8 mg per day (mg/day) was continued for the remaining period of treatment."
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Started | 361 | 179 | 180
Full Analysis Set (FAS) | 361 | 179 | 180
Safety Analysis Set (SAS) | 358 | 175 | 180
Exposed | 358 | 175 | 180
Completed | 341 | 167 | 151
Not Completed | 20 | 12 | 29
Not completed — Adverse Event | 5 | 1 | 15
Not completed — Protocol Violation | 3 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 10 | 8 | 8
Not completed — Severe hypoglycaemic episode | 0 | 0 | 1
Not completed — Non-compliance towards treatment | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS included all randomised participants.
Groups:
- Insulin Degludec/Liraglutide: Participants were to receive Insulin degludec/liraglutide subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 10 dose steps (10 units insulin degludec and 0.36 mg liraglutide) initially. The dose was then adjusted twice weekly based on pre-breakfast self-measured plasma glucose (SMPG) target of 4.0-5.0 mmol/L. The maximum dose was 50 dose steps (50 units insulin degludec and 1.8 mg liraglutide). One dose step corresponded to 1 unit insulin degludec per 0.036 mg liraglutide.
- Liraglutide: Participants were to receive liraglutide subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 0.6 mg initially. The dose was then escalated in weekly increments of 0.6 mg to reach a target dose of 1.8 mg. Liraglutide dose of 1.8 mg/day was continued for the remaining period of treatment."
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide | Total
Number analyzed (Participants) | 361 | 179 | 180 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.3) | 55.7 (10.2) | 54.1 (10.2) | 54.7 (10.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 142 | 79 | 72 | 293
  Male | 219 | 100 | 108 | 427
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 361 | 179 | 180 | 720
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 361 | 179 | 180 | 720
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage points of HbA1c] | 8.20 (0.83) | 8.31 (0.84) | 8.21 (0.77) | 8.23 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in HbA1c from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage points of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Percentage points of HbA1c | -1.71 (0.88) | -1.20 (0.99) | -1.16 (0.89)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The change from baseline in HbA1c after 26 weeks of treatment was analysed using an analysis of covariance (ANCOVA) model with treatment and previous oral anti-diabetic (OAD) treatment as fixed factors and baseline HbA1c as covariate. Missing values were imputed by last observation carried forward (LOCF); Test type: Non-Inferiority — Non-inferiority of insulin degludec/liraglutide versus insulin degludec was considered as confirmed if the 95% confidence interval (CI) for the mean treatment difference lied entirely below 0.4%. Non-inferiority was investigated on the FAS; p < 0.0001, ANCOVA; Mean treatment difference = -0.59, 95% CI 2-sided [-0.73 to -0.46]
Statistical Analysis 2: Comparison: Insulin Degludec/Liraglutide vs Liraglutide; The change from baseline in HbA1c after 26 weeks of treatment was analysed using an ANCOVA model with treatment and previous OAD treatment as fixed factors and baseline HbA1c as covariate. Missing values were imputed by LOCF; Test type: Superiority; p < 0.0001, ANCOVA; Mean treatment difference = -0.63, 95% CI 2-sided [-0.76 to -0.49]

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Kilogram (Kg) | 0.2 (2.7) | 1.3 (2.7) | -2.5 (2.7)

3. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification (requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or blood glucose (BG) confirmed by a plasma glucose (PG) value < 3.1 millimoles per liter (mmol/L) with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. The number of episodes are represented as rates. The observed rates of treatment-emergent severe or BG confirmed hypoglycaemic episodes per patient years of exposure (PYE) (number of episodes divided by PYE multiplied by 100) during 26 weeks of treatment are presented.
Time Frame: Weeks 0-26
Population: Safety analysis set (SAS) included all participants who received at least one dose of insulin degludec/liraglutide, insulin degludec or liraglutide. Overall number of participants analysed = number of participants with available data.
Measure: Number; unit: (Number of episodes/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 29 | 14 | 3
(Number of episodes/PYE)*100 | 23.94 | 17.01 | 3.60

4. Secondary Outcome: Insulin Dose
Description: The actual daily total insulin dose after 26 weeks of treatment is presented. This outcome measure is only applicable for Insulin degludec/liraglutide and Insulin degludec treatment arms.
Time Frame: Week 26
Population: SAS included all participants receiving at least one dose of the insulin degludec/liraglutide or insulin degludec. Overall number of participants analysed = participants with available data
Measure: Mean (Standard Deviation); unit: Units of insulin (U)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 340 | 167
Units of insulin (U) | 24.8 (11.9) | 30.1 (14.4)

5. Secondary Outcome: Participants Who Achieved HbA1c < 7.0%, American Diabetes Association (ADA) Target (Yes/no)
Description: Number of participants who achieved ADA HbA1c target (HbA1c < 7.0%) (yes/no) after 26 weeks of treatment are presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysied = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Participants
  Yes | 272 | 83 | 80
  No | 69 | 84 | 71

6. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5%, International Diabetes Federation (IDF) Target (Yes/no)
Description: Number of participants who achieved IDF HbA1c target (HbA1c ≤ 6.5%) (yes/no) after 26 weeks of treatment are presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Participants
  Yes | 201 | 48 | 41
  No | 140 | 119 | 110

7. Secondary Outcome: Participants Who Achieved HbA1c <7.0% and Change in Body Weight From Baseline Below or Equal to Zero
Description: Number of participants who achieved ADA HbA1c target (HbA1c < 7.0%) (yes/no) and change from baseline in body weight below or equal to zero after 26 weeks are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 147 | 34 | 74
  No | 214 | 145 | 106

8. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% and Change From Baseline in Body Weight Below or Equal to Zero
Description: Number of participants who achieved IDF HbA1c target (HbA1c ≤ 6.5%) (yes/no) and change from baseline in body weight below or equal to zero after 26 weeks are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 111 | 21 | 37
  No | 250 | 158 | 143

9. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% Without Severe or Blood Glucose (BG) Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of participants who achieved ADA HbA1c target (HbA1c <7.0%) (yes/no) after 26 weeks of treatment and without severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 265 | 80 | 84
  No | 96 | 99 | 96

10. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% Without Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of participants who achieved IDF HbA1c target (HbA1c ≤ 6.5%) (yes/no) after 26 weeks of treatment and without severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 195 | 46 | 43
  No | 166 | 133 | 137

11. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% Without Severe or BG Confirmed Episodes, and Change From Baseline in Body Weight Below or Equal to Zero.
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of participants who achieved ADA HbA1c target (HbA1c < 7.0%) (yes/no) after 26 weeks of treatment without severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment and with change from baseline in body weight below or equal to zero are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 136 | 33 | 72
  No | 225 | 146 | 108

12. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% Without Severe or BG Confirmed Episodes and Change From Baseline in Body Weight Below or Equal to Zero.
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of participants who achieved IDF HbA1c target (HbA1c ≤ 6.5%) (yes/no) after 26 weeks of treatment without severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment and with change from baseline in body weight below or equal to zero are presented. Missing values are imputed by LOCF.
Time Frame: Week 26
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
Participants
  Yes | 103 | 21 | 36
  No | 258 | 158 | 144

13. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
mmol/L | -3.64 (2.27) | -3.45 (2.34) | -1.86 (2.11)

14. Secondary Outcome: Change in Waist Circumferance
Description: Change from baseline (week 0) in waist circumferance after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 166 | 151
Centimeters (cm) | -0.3 (3.4) | 1.2 (4.2) | -2.6 (3.8)

15. Secondary Outcome: 9-point SMPG Profile
Description: Participants measured their PG levels using blood glucose meters at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). 9-point SMPG values at 26 weeks of treatment are presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Number analysed= number of participants with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 361 | 179 | 180
mmol/L
  Before breakfast: number analyzed (Participants) | 337 | 165 | 151
  Before breakfast | 5.41 (1.07) | 5.66 (1.20) | 6.89 (1.37)
  90 minutes after the start of breakfast: number analyzed (Participants) | 336 | 161 | 151
  90 minutes after the start of breakfast | 8.97 (2.48) | 9.85 (2.73) | 10.04 (2.81)
  Before lunch: number analyzed (Participants) | 334 | 162 | 151
  Before lunch | 6.31 (1.80) | 7.10 (2.35) | 7.48 (2.14)
  90 minutes after the start of the lunch: number analyzed (Participants) | 334 | 161 | 151
  90 minutes after the start of the lunch | 8.87 (2.15) | 10.18 (2.81) | 9.54 (2.43)
  Before dinner: number analyzed (Participants) | 335 | 164 | 151
  Before dinner | 6.52 (1.77) | 7.39 (2.23) | 7.50 (2.11)
  90 minutes after start of the dinner: number analyzed (Participants) | 332 | 164 | 151
  90 minutes after start of the dinner | 9.33 (2.40) | 10.27 (2.68) | 9.45 (2.13)
  At bedtime: number analyzed (Participants) | 330 | 160 | 150
  At bedtime | 7.99 (2.28) | 8.86 (2.38) | 8.49 (2.26)
  At 4:00 am: number analyzed (Participants) | 326 | 158 | 148
  At 4:00 am | 5.60 (1.26) | 6.12 (1.75) | 6.86 (1.60)
  Before breakfast the following day: number analyzed (Participants) | 336 | 165 | 150
  Before breakfast the following day | 5.35 (0.96) | 5.47 (1.07) | 6.81 (1.47)

16. Secondary Outcome: Change in Mean of 9-point SMPG Profile
Description: Participants measured their PG levels using blood glucose meters at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). The mean of profile is defined as the area under the profile divided by measurement time and is calculated using the trapezoidal method. Change in mean of the 9-point SMPG profile from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 331 | 162 | 146
mmol/L | -3.17 (2.16) | -2.47 (2.14) | -2.13 (2.02)

17. Secondary Outcome: Change in Mean Post-prandial Plasma Glucose (PG) Increments
Description: Participants measured their PG levels using blood glucose meters at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). Post-prandial SMPG increments from before meal to 90 minutes after for breakfast, lunch and dinner were calculated. The mean increment over all meals was derived as the mean of all available meal increments. Change from baseline (week 0) in post-prandial SMPG increments for all meals after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 335 | 164 | 150
mmol/L | -0.20 (2.40) | 0.09 (2.40) | -0.54 (2.57)

18. Secondary Outcome: Change in Fasting C-peptide - Ratio to Baseline
Description: Change in fasting C-peptide (measured in nanomoles per liter [nmol/L]) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall, number of participants analysed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting C-peptide
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 339 | 167 | 150
Ratio of fasting C-peptide | 0.54 (52.8) | 0.38 (68.5) | 0.98 (37.6)

19. Secondary Outcome: Change in Fasting Human Insulin - Ratio to Baseline
Description: Change in fasting human insulin (measured in picomoles per liter [pmol/L]) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting human insulin
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 328 | 162 | 142
Ratio of fasting human insulin | 0.53 (71.7) | 0.38 (77.6) | 1.04 (53.3)

20. Secondary Outcome: Change in Fasting Glucagon - Ratio to Baseline
Description: Change in fasting glucagon (measured in picograms per milliliter [pg/mL]) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of particiapants analysed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting glucagon
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 338 | 165 | 150
Ratio of fasting glucagon | 0.90 (76.6) | 0.95 (56.4) | 0.98 (75.9)

21. Secondary Outcome: Change in HOMA-B (Beta Cell Function)- Ratio to Baseline
Description: Change in HOMA-B (measured in %) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-B (beta cell function)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 328 | 162 | 141
Ratio of HOMA-B (beta cell function) | 1.38 (77.3) | 0.94 (77.4) | 1.53 (63.8)

22. Secondary Outcome: Change in Fasting Total Cholesterol - Ratio to Baseline
Description: Change in fasting total cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Ratio of fasting total cholesterol | 0.94 (19.1) | 0.99 (16.8) | 0.97 (17.7)

23. Secondary Outcome: Change in Fasting High Density Lipoprotein (HDL) Cholesterol- Ratio to Baseline
Description: Change in fasting HDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Ratio of fasting HDL cholesterol | 1.01 (14.7) | 1.02 (15.7) | 1.03 (14.8)

24. Secondary Outcome: Change in Fasting Low Density Lipoprotein (LDL) Cholesterol- Ratio to Baseline
Description: Change in fasting LDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 340 | 167 | 151
Ratio of fasting LDL cholesterol | 0.92 (34.2) | 1.01 (36.2) | 0.96 (34.4)

25. Secondary Outcome: Change in Fasting Very Low-density Lipoprotein (VLDL) Cholesterol- Ratio to Baseline
Description: Change in fasting VLDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting VLDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Ratio of fasting VLDL cholesterol | 0.90 (49.9) | 0.84 (47.2) | 0.92 (38.6)

26. Secondary Outcome: Change in Fasting Triglycerides - Ratio to Baseline.
Description: Change in fasting triglycerides (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Ratio of fasting triglycerides | 0.88 (54.4) | 0.82 (50.5) | 0.90 (45.2)

27. Secondary Outcome: Change in Fasting Free Fatty Acid - Ratio to Baseline
Description: Change in fasting free fatty acid (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting free fatty acid
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 340 | 167 | 150
Ratio of fasting free fatty acid | 0.55 (69.9) | 0.48 (76.5) | 0.80 (69.3)

28. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAE)
Description: A TEAE was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. The observed rates of adverse events (AEs) per patient years of exposure (PYE) (number of AEs divided by PYE multiplied by 100) after 26 weeks are presented.
Time Frame: Weeks 0-26
Population: SAS included all participants who received at least one dose of Insulin degludec/liraglutide, insulin degludec or liraglutide. Number of participants analysed = number of participants with available data.
Measure: Number; unit: (Number of AEs/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 267 | 117 | 143
(Number of AEs/PYE)*100 | 410.82 | 306.19 | 541.00

29. Secondary Outcome: Number of Treatment Emergent Nocturnal Severe or BG Confirmed Hypoglycaemic Episodes.
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Hypoglycaemic episodes were defined as nocturnal if the time of the onset was between 00:01 and 05.59 both inclusive. The number of episodes are represented as rates. The observed rates of episodes per PYE (number of episodes divided by PYE multiplied by 100) after 26 weeks of treatment are presented.
Time Frame: Weeks 0-26
Population: SAS included all participants who received at least one dose of insulin degludec/liraglutide, insulin degludec or liraglutide. Overall number of participants analysed = number of participants with available data.
Measure: Number; unit: (Number of episodes/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 6 | 4 | 0
(Number of episodes/PYE)*100 | 4.45 | 4.54 |

30. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes.
Description: Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. The number of episodes are represented as rates. The observed rates of episodes per PYE (number of episodes divided by PYE multiplied by 100) after 26 weeks of treatment are presented.
Time Frame: Weeks 0-26
Population: as for outcome 29
Measure: Number; unit: (Number of episodes/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 20 | 8 | 1
(Number of episodes/PYE)*100 | 15.03 | 9.07 | 1.20

31. Secondary Outcome: Number of Treatment Emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Hypoglycaemic episodes were defined as nocturnal if the time of the onset was between 00:01 and 05.59 both inclusive. The number of episodes are represented as rates. The observed rates of episodes per PYE (number of episodes divided by PYE multiplied by 100) after 26 weeks of treatment are presented.
Time Frame: Weeks 0-26
Population: as for outcome 29
Measure: Number; unit: (Number of episodes/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 5 | 3 | 0
(Number of episodes/PYE)*100 | 2.78 | 3.40 |

32. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to ADA Definition
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. The number of episodes are represented as rates. The observed rates of episodes (according to the ADA definition) per PYE (number of episodes divided by PYE multiplied by 100) after 26 weeks of treatment are presented.
Time Frame: Weeks 0-26
Population: as for outcome 29
Measure: Number; unit: (Number of episodes/PYE)*100
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 236 | 123 | 19
(Number of episodes/PYE)*100 | 668.55 | 746.20 | 37.19

33. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as cardiovascular system; central and peripheral nervous system; gastrointestinal system including mouth; general appearance; head, ears, eyes, nose, throat, neck; lymph node palpation; musculoskeletal system; respiratory system; skin and thyroid gland. The number of participants assessed as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) at screening (week -2) and week 26 per each category is presented.
Time Frame: Week -2, week 26
Population: SAS included all participants who received at least one dose of Insulin degludec/liraglutide, insulin degludec or liraglutide. Overall number of participants analyzed=participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 358 | 175 | 180
Participants
  Week -2: Cardiovascular system: Normal | 353 | 173 | 180
  Week -2: Cardiovascular system: Abnormal, NCS | 2 | 2 | 0
  Week -2: Cardiovascular system: Abnormal CS | 3 | 0 | 0
  Week 26: Cardiovascular system: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Cardiovascular system: Normal | 336 | 166 | 151
  Week 26: Cardiovascular system: Abnormal, NCS | 3 | 1 | 0
  Week 26: Cardiovascular system: Abnormal CS | 2 | 0 | 0
  Week -2: Central and peripheral nervous system: Normal | 355 | 172 | 179
  Week -2: Central and peripheral nervous system: Abnormal, NCS | 1 | 0 | 0
  Week -2: Central and peripheral nervous system: Abnormal CS | 2 | 3 | 1
  Week 26: Central and peripheral nervous system: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Central and peripheral nervous system: Normal | 338 | 164 | 150
  Week 26: Central and peripheral nervous system: Abnormal, NCS | 1 | 0 | 0
  Week 26: Central and peripheral nervous system: Abnormal CS | 2 | 3 | 1
  Week -2: Gastrointestinal system including mouth: Normal | 355 | 174 | 179
  Week -2: Gastrointestinal system including mouth: Abnormal, NCS | 3 | 1 | 1
  Week -2: Gastrointestinal system including mouth: Abnormal CS | 0 | 0 | 0
  Week 26: Gastrointestinal system including mouth: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Gastrointestinal system including mouth: Normal | 339 | 166 | 150
  Week 26: Gastrointestinal system including mouth: Abnormal, NCS | 2 | 1 | 1
  Week 26: Gastrointestinal system including mouth: Abnormal CS | 0 | 0 | 0
  Week -2: General appearance: Normal | 351 | 169 | 177
  Week -2: General appearance: Abnormal, NCS | 3 | 2 | 1
  Week -2: General appearance: Abnormal CS | 4 | 4 | 2
  Week 26: General appearance: number analyzed (Participants) | 341 | 167 | 151
  Week 26: General appearance: Normal | 336 | 161 | 150
  Week 26: General appearance: Abnormal, NCS | 2 | 2 | 0
  Week 26: General appearance: Abnormal CS | 3 | 4 | 1
  Week -2: Head, ears, eyes, nose, throat, neck: Normal | 348 | 170 | 175
  Week -2: Head, ears, eyes, nose, throat, neck: Abnormal, NCS | 6 | 4 | 3
  Week -2: Head, ears, eyes, nose, throat, neck: Abnormal CS | 4 | 1 | 2
  Week 26: Head, ears, eyes, nose, throat, neck: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Head, ears, eyes, nose, throat, neck: Normal | 332 | 164 | 150
  Week 26: Head, ears, eyes, nose, throat, neck: Abnormal, NCS | 6 | 3 | 1
  Week 26: Head, ears, eyes, nose, throat, neck: Abnormal CS | 3 | 0 | 0
  Week -2: Lymph node palpation: Normal | 357 | 174 | 180
  Week -2: Lymph node palpation: Abnormal, NCS | 0 | 0 | 0
  Week -2: Lymph node palpation: Abnormal CS | 1 | 1 | 0
  Week 26: Lymph node palpation: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Lymph node palpation: Normal | 340 | 166 | 151
  Week 26: Lymph node palpation: Abnormal, NCS | 0 | 0 | 0
  Week 26: Lymph node palpation: Abnormal CS | 1 | 1 | 0
  Week -2: Musculoskeletal system: Normal | 353 | 172 | 177
  Week -2: Musculoskeletal system: Abnormal, NCS | 2 | 2 | 0
  Week -2: Musculoskeletal system: Abnormal CS | 3 | 1 | 3
  Week 26: Musculoskeletal system: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Musculoskeletal system: Normal | 332 | 165 | 149
  Week 26: Musculoskeletal system: Abnormal, NCS | 2 | 1 | 0
  Week 26: Musculoskeletal system: Abnormal CS | 7 | 1 | 2
  Week-2: Respiratory system: Normal | 358 | 175 | 180
  Week-2: Respiratory system: Abnormal, NCS | 0 | 0 | 0
  Week-2: Respiratory system: Abnormal CS | 0 | 0 | 0
  Week 26: Respiratory system: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Respiratory system: Normal | 341 | 167 | 151
  Week 26: Respiratory system: Abnormal, NCS | 0 | 0 | 0
  Week 26: Respiratory system: Abnormal CS | 0 | 0 | 0
  week -2: Skin: Normal | 312 | 152 | 156
  week -2: Skin: Abnormal, NCS | 37 | 20 | 20
  week -2: Skin: Abnormal CS | 9 | 3 | 4
  Week 26: Skin: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Skin: Normal | 297 | 146 | 134
  Week 26: Skin: Abnormal, NCS | 36 | 19 | 15
  Week 26: Skin: Abnormal CS | 8 | 2 | 2
  Week -2: Thyroid gland: Normal | 348 | 171 | 179
  Week -2: Thyroid gland: Abnormal, NCS | 5 | 1 | 1
  Week -2: Thyroid gland: Abnormal CS | 5 | 3 | 0
  Week 26: Thyroid gland: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Thyroid gland: Normal | 334 | 163 | 151
  Week 26: Thyroid gland: Abnormal, NCS | 3 | 2 | 0
  Week 26: Thyroid gland: Abnormal CS | 4 | 2 | 0

34. Secondary Outcome: Eye Examination
Description: Dilated fundoscopy or fundus photography was performed by the investigator at screening (week -2) and week 26. The results of the examination were interpreted for each eye (left and right) and are categorised as normal, abnormal NCS or abnormal CS. Number of participants in each category at screening (week -2) and week 26 is presented.
Time Frame: Week -2, Week 26
Population: SAS included all participants who received at least one dose of insulin degludec/liraglutide, insulin degludec or liraglutide. Overall number of participants analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 358 | 175 | 180
Participants
  Week -2: Left eye: Normal | 222 | 109 | 110
  Week -2: Left eye: Abnormal, NCS | 45 | 14 | 20
  Week -2: Left eye: Abnormal, CS | 91 | 52 | 50
  Week 26: Left eye: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Left eye: Normal | 217 | 99 | 100
  Week 26: Left eye: Abnormal, NCS | 39 | 20 | 13
  Week 26: Left eye: Abnormal, CS | 85 | 48 | 38
  Week -2: Right eye: Normal | 230 | 112 | 111
  Week -2: Right eye: Abnormal, NCS | 42 | 16 | 22
  Week -2: Right eye: Abnormal, CS | 86 | 47 | 47
  Week 26: Right eye: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Right eye: Normal | 217 | 103 | 96
  Week 26: Right eye: Abnormal, NCS | 40 | 23 | 15
  Week 26: Right eye: Abnormal, CS | 84 | 41 | 40

35. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: Electrocardiogram was assessed by the investigator as normal, abnormal NCS and abnormal CS. Number of participants at screening (week -2) and at week 26 is presented.
Time Frame: Week -2, week 26
Population: SAS included all participants who received at least one dose of insulin degludec/liraglutide, insulin degludec or liraglutide. Number of participants analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 358 | 175 | 180
Participants
  Week -2: Normal | 223 | 109 | 108
  Week -2: Abnormal, NCS | 94 | 46 | 52
  Week -2: Abnormal CS | 41 | 20 | 20
  Week 26: number analyzed (Participants) | 341 | 167 | 151
  Week 26: Normal | 227 | 108 | 87
  Week 26: Abnormal, NCS | 76 | 47 | 40
  Week 26: Abnormal CS | 38 | 12 | 24

36. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline (week 0) after 26 weeks of treatment is presented
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Beats per minuts (beats/min)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Beats per minuts (beats/min) | 4.6 (8.6) | -0.1 (8.6) | 4.9 (9.7)

37. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change in blood pressure (systolic and diastolic blood pressure) from baseline (week 0) after 26 weeks of treatment is presented
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3.5 (12.7) | -1.2 (11.7) | -3.3 (13.8)
  Distolic blood pressure | -0.4 (8.3) | -0.7 (8.1) | 0.0 (8.4)

38. Secondary Outcome: Change in Biochemistry Parameters: Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase, Amalyse, Lipase, Creatiine Kinase Serum
Description: Change in alkaline phosphatase, ALT, AST, creatine kinase, amylase, lipase, creatine kinase serum from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
Units per liter (U/L)
  Alkaline phosphatase | -2.0 (14.85) | -2.29 (11.49) | -0.48 (14.11)
  ALT | -4.63 (13.06) | -6.17 (13.54) | -2.81 (16.97)
  AST | -1.31 (7.94) | -2.65 (8.40) | -0.99 (9.64)
  Creatine kinase | 10.67 (100.87) | 15.37 (52.99) | 0.52 (56.20)
  Amylase | 9.84 (36.73) | 5.09 (14.68) | 5.68 (13.70)
  Lipase | 16.13 (101.19) | -1.87 (15.64) | 14.11 (19.76)

39. Secondary Outcome: Change in Biochemistry Parameters (Albumin Serum, Total Protein)
Description: Change in total protein, albumin serum from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: grams per decileter (g/dL)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
grams per decileter (g/dL)
  Albumin serum | -0.05 (0.28) | -0.09 (0.26) | 0.04 (0.26)
  Total protein | -0.08 (0.42) | -0.08 (0.39) | -0.01 (0.39)

40. Secondary Outcome: Change in Biochemistry Parameters: Calcium Serum (Total), Calcium Corrected Serum, Potassium Serum, Sodium Serum, Urea Serum
Description: Change in calcium serum (total), calcium corrected serum, potassium serum, sodium serum, urea serum from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
mmol/L
  Calcium serum (total) | -0.01 (0.10) | -0.02 (0.10) | -0.00 (0.09)
  Calcium corrected serum | -0.00 (0.08) | -0.00 (0.08) | -0.01 (0.07)
  Sodium serum | 1.21 (2.09) | 0.98 (2.37) | 0.32 (2.12)
  Urea serum | 0.05 (0.57) | 0.03 (0.53) | 0.16 (0.67)
  Potassium serum | -0.04 (0.34) | -0.09 (0.39) | -0.04 (0.34)

41. Secondary Outcome: Change in Biochemistry Parameters: Total Bilirubin Serum, Creatinine Serum
Description: Change in total bilirubin serum, creatinine serum from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 151
micromoles per liter (umol/L)
  Total bilirubin | -0.78 (3.35) | -0.55 (4.52) | -1.16 (3.92)
  creatinine serum | 1.02 (8.41) | 1.36 (7.92) | -0.60 (7.89)

42. Secondary Outcome: Change in Haematological Parameter: Erythrocytes Blood
Description: Change in erythrocyte blood from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
10^12 cells per liter (10^12/L) | -0.05 (0.27) | -0.00 (0.27) | -0.05 (0.25)

43. Secondary Outcome: Change in Haematological Parameter: Haematocrits
Description: Change in haematocrits from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage points (%) of red blood cells
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
Percentage points (%) of red blood cells | -0.56 (2.65) | -0.49 (2.69) | -0.42 (2.57)

44. Secondary Outcome: Change in Haemotological Parameter- Eosinophils
Description: Change in eosinophils from baseline after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: % of eosinophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
% of eosinophils | -0.06 (1.90) | 0.19 (1.73) | 0.11 (1.94)

45. Secondary Outcome: Change in Haematological Parameter - Neutrophils
Description: Change in neutrophils from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: % of neutrophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
% of neutrophils | 0.57 (6.46) | 0.18 (7.70) | -0.53 (7.05)

46. Secondary Outcome: Change in Haematological Parameter: Basophils
Description: Change in basophils from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: % of basophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
% of basophils | -0.02 (0.29) | -0.01 (0.28) | -0.03 (0.26)

47. Secondary Outcome: Change in Haemotological Parameter- Monocytes
Description: Change in monocytes from baseline (week 0) after 26 weeks of treatment is presented
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: % of monocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
% of monocytes | -0.03 (1.92) | 0.01 (1.85) | 0.05 (2.13)

48. Secondary Outcome: Change in Haematological Parameter - Lymphocytes
Description: Change in lymphocytes from baseline (week 0) after 26 weeks of treatment is presented
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: % of lymphocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
% of lymphocytes | -0.46 (6.04) | -0.38 (7.12) | 0.40 (6.11)

49. Secondary Outcome: Change in Haematology: Haemoglobin Blood
Description: Change in haemoglobin from baseline (week 0) after 26 weeks of treatment is presented.
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
mmol/L | -0.10 (0.53) | -0.06 (0.48) | -0.05 (0.47)

50. Secondary Outcome: Change in Haematologcal Parameter: Leukocytes
Description: Change in leukocytes from baseline (week 0) after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 341 | 167 | 150
10^9 cells per liter (10^9/L) | 0.25 (1.18) | 0.23 (1.41) | -0.01 (1.14)

51. Secondary Outcome: Change in Haematological Parameter: Thrombocytes
Description: Change in thrombocytes from baseline (week 0) after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 340 | 167 | 149
10^9 cells per liter (10^9/L) | 8.19 (28.02) | 8.32 (34.48) | 4.32 (33.39)

52. Secondary Outcome: Change in Calcitonin
Description: Calcitonin levels were measured and were categorised as low, normal or high in relation to reference range (8.31- 14.3 picogram/milliliter [pg/mL]). Number of participants in each category at baseline (week 0) and week 26 are presented.
Time Frame: Week 0, week 26
Population: SAS included all participants who received at least one dose of Insulin degludec/liraglutide, insulin degludec or liraglutide. Number analysed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 358 | 175 | 180
Participants
  Week 0: Low | 0 | 0 | 0
  Week 0: Normal | 351 | 172 | 178
  Week 0: High | 7 | 3 | 2
  Week 26: number analyzed (Participants) | 340 | 167 | 150
  Week 26: Low | 0 | 0 | 0
  Week 26: Normal | 334 | 165 | 147
  Week 26: High | 6 | 2 | 3

53. Secondary Outcome: Urinalysis (Protein, Glucose, Erythrocytes and Ketones)
Description: The urinalysis assessment was the measurements of protein, glucose, erythrocytes and ketones in urine at baseline (week 0) and week 26 and categorised as negative, trace and positive. Number of participants in each category at week 0 and week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 357 | 175 | 180
Participants
  Week 0: Erythrocytes: Negative | 299 | 153 | 156
  Week 0: Erythrocytes: Trace | 36 | 16 | 16
  Week 0: Erythrocytes: Positive | 22 | 6 | 8
  Week 26: Erythrocytes: number analyzed (Participants) | 339 | 167 | 151
  Week 26: Erythrocytes: Negative | 297 | 146 | 136
  Week 26: Erythrocytes: Trace | 28 | 16 | 11
  Week 26: Erythrocytes: Positive | 14 | 5 | 4
  Week 0: Glucose: Negative | 253 | 119 | 123
  Week 0: Glucose: Trace | 35 | 19 | 18
  Week 0: Glucose: Positive | 69 | 37 | 39
  Week 26: Glucose: number analyzed (Participants) | 339 | 167 | 151
  Week 26: Glucose: Negative | 322 | 157 | 131
  Week 26: Glucose: Trace | 11 | 3 | 5
  Week 26: Glucose: Positive | 6 | 7 | 15
  Week 0: Ketones: Negative | 325 | 152 | 167
  Week 0: Ketones: Trace | 25 | 20 | 11
  Week 0: Ketones: Positive | 7 | 3 | 2
  Week 26: Ketones: number analyzed (Participants) | 339 | 167 | 151
  Week 26: Ketones: Negative | 334 | 163 | 141
  Week 26: Ketones: Trace | 4 | 3 | 10
  Week 26: Ketones: Positive | 1 | 1 | 0
  Week 0: Protein: Negative | 216 | 104 | 116
  Week 0: Protein: Trace | 86 | 40 | 37
  Week 0: Protein: Positive | 55 | 31 | 27
  Week 26: Protein: number analyzed (Participants) | 339 | 167 | 151
  Week 26: Protein: Negative | 254 | 120 | 105
  Week 26: Protein: Trace | 58 | 26 | 28
  Week 26: Protein: Positive | 27 | 21 | 18

54. Secondary Outcome: Occurence of Anti-insulin Degludec Specific Antibodies
Description: This outcome measure is only applicable for the insulin degludec/liraglutide arm and insulin degludec arm. Serum samples were analysed for the presence of anti-insulin degludec specific antibodies. Results at week 27 are presented as percentage of bound radioactive-labelled insulin (B) /total radioactive-labelled insulin added to the samples (T).
Time Frame: Week 27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 332 | 166
%B/T | 0.22 (1.02) | 0.12 (0.79)

55. Secondary Outcome: Occurence of Antibodies Cross-reacting to Human Insulin
Description: This outcome measure is only applicable for the insulin degludec/liraglutide arm and insulin degludec arm. Serum samples were analysed for the presence of cross-reacting antibodies to human insulin. Results at week 27 are presented as percentage of bound radioactive-labelled insulin (B) /total radioactive-labelled insulin added to the samples (T).
Time Frame: Week 27
Population: SAS included all participants who received at least one dose of insulin degludec/liraglutide or insulin degludec. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 332 | 166
%B/T | 6.61 (15.00) | 2.99 (10.89)

56. Secondary Outcome: Occurence of Total Insulin Antibodies
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide arm and Insulin degludec arm. Serum samples were analysed for the presence of antobodies to human insulin. Results at week 27 are presented as percentage of bound radioactive-labelled insulin (B) /total radioactive-labelled insulin added to the samples (T).
Time Frame: Week 27
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 332 | 166
%B/T | 6.83 (15.78) | 3.11 (11.42)

57. Secondary Outcome: Occurence of Anti-liraglutide Antibodies
Description: This outcome measure is applicable for the Insulin degludec/liraglutide arm and the liraglutide arm. Serum samples were analysed for the presence of anti-liraglutide antibodies. Number of participants who were assessed for anti-liraglutide antibodies at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 55
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 332 | 160
Participants
  Yes | 45 | 40
  No | 287 | 120

58. Secondary Outcome: Occurence of Antibodies Cross-reacting to Native Glucagon-like Peptide (GLP-1)
Description: This outcome measure is applicable to the Insulin degludec/liraglutide arm and the liraglutide arm. Serum samples were analysed for the presence of cross-reacting antibodies to native GLP-1. Number of participants who measured with anti-liraglutide antibodies cross reacting native GLP-1 at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 55
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 332 | 160
Participants | 6 | 3

59. Secondary Outcome: Occurence of Neutralising Liraglutide Antibodies
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide arm and liraglutide arm. Neutralising antibodies were assessed when the corresponding anti-Liraglutide antibody were positive at week 27. Number of participants who measured with neutralising liraglutide antibodies at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 332 | 160
Participants | 9 | 8

60. Secondary Outcome: Occurence of Neutralising Antibodies Cross-reacting to Native GLP-1
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide arm and liraglutide arm. Cross reacting antibodies were assessed when anti-liraglutide antibody was positive. Number of participants who measured with neutralising liraglutide antibodies cross-reacting to native GLP-1 at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 332 | 160
Participants | 0 | 0

61. Secondary Outcome: Serum Concentrations of Insulin Degludec
Description: This outcome measure is applicable for Insulin degludec and Insulin degludec/liraglutide arms. Serum samples from the Insulin degludec/liraglutide and Insulin degludec arms were assayed using population PK analysis. The maximum serum concentrations (Cmax) are summarised for the two arms.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall the number of participants analysed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 339 | 168
pmol/L | 3583 (55.9) | 4133 (52.8)

62. Secondary Outcome: Plasma Concentration of Liraglutide
Description: This outcome measure is for Insulin degludec/liraglutide and liraglutide arms. Serum samples from the Insulin degludec/liraglutide and liraglutide arms were assayed using population PK analysis. The Cmax are summarised for the two arms.
Time Frame: Week 0, week 26
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 339 | 165
pmol/L | 9963 (50.4) | 21602 (37)

ADVERSE EVENTS:
Time Frame: Weeks 0-30
Description: A TEAE was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. Results are based on SAS which included all participants who received at least one dose of insulin degludec/liraglutide, insulin degludec or liraglutide
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/358 | 0/175 | 0/180
Serious Adverse Events (participants affected / at risk) | 14/358 | 7/175 | 14/180
Other Adverse Events (participants affected / at risk) | 161/358 | 55/175 | 98/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=358) | Insulin Degludec (N=175) | Liraglutide (N=180)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mass excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=358) | Insulin Degludec (N=175) | Liraglutide (N=180)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 2 (2) | 26 (27)
Diabetic retinopathy (Eye disorders) | 28 (28) | 6 (6) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 23 (31) | 3 (3) | 26 (41)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 10 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 16 (16) | 6 (6) | 10 (11)
Lipase increased (Investigations) | 27 (30) | 5 (6) | 22 (22)
Nasopharyngitis (Infections and infestations) | 16 (20) | 9 (11) | 5 (7)
Nausea (Gastrointestinal disorders) | 14 (25) | 1 (1) | 21 (23)
Upper respiratory tract infection (Infections and infestations) | 66 (83) | 31 (34) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03172494/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03172494/SAP_001.pdf